CLINICAL TRIAL: NCT04334473
Title: Intraocular Pressure and Ocular Biometrics Changes After Phacoemulsification in Glaucomatous Patients and Age Matched Controls, Comparative Study
Brief Title: IOP and Ocular Biometrics Changes After Phacoemulsification in Glaucoma Patients and Controls
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mai Nasser Abd Elmohsen (Other)
Responsible Party: Sponsor-Investigator, Mai Nasser Abd Elmohsen, Lecturer of ophthalmology, Kasr El Aini Hospital
Organization: Kasr El Aini Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: N-45-2019
Record Dates: First submitted 2020-04-02; First posted 2020-04-06 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Glaucoma; Cataract
Keywords: Ocular bio-metrics; Anterior chamber depth; UBM
MeSH Terms: conditions — Glaucoma; Cataract | interventions — Phacoemulsification; Lens Implantation, Intraocular

STUDY DESIGN:
Intervention Model Description: All participants are assigned to the same interventions. All will undergo pre- & postoperative assessment, cataract surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cataract patients (Other): Patients having cataract candidates for phacoemulsification with or without glaucoma are prepared to do cataract surgery with preoperative and postoperative assessment of intraocular pressure and ocular bio-metrics using UBM.
  Interventions: Procedure: phacoemulsification and Intraocular lens implantation; Diagnostic Test: Ultrasound Biomicrosopy (UBM)

INTERVENTIONS:
Procedure: phacoemulsification and Intraocular lens implantation — Standartd surgical procedure with small incision to remove catarct using ultrasound waves. it can be done by topica, local or general anaesthesia acoording to patients general fitness and preference.
Diagnostic Test: Ultrasound Biomicrosopy (UBM) — A diagnostic test using ultrasound waves to evaluate the anterior chamber depth, angle and lens vault.

SUMMARY:
Effect of phacoemulsification on intraocular pressure has been studied with variable results.Furthermore, effect of phacoemulsification on ocular biometrics including anterior chamber depth and angle opening distance has also been studied. In our study we aim at establishing a quantitative relationship between preoperative ocular biometrics and postoperative intraocular pressure change and comparing this relationship in glaucomatous and non-glaucomatous eyes.

DETAILED DESCRIPTION:
All patients will have the anterior chamber angle assessed by indentation gonioscopy preoperatively. Anterior Chamber Depth & lens thickness will be measured by Optical Biometry (lenstar 900) as well as measurement of the angle & lens vault using the Ultrasound Biomicrosopy (UBM) before and 1 month after cataract surgery. IOP will be measured pre- & postoperatively on day 7 and 30. Possible Risk (s): Risks of surgery(hemorrhage, endophthalmitis), Risks for investigations: minimal risk of infection To minimize the risk of infection: adherence to pre-& intraoperative infection-control measures, postoperative UBM is to be done at 1 month.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-70 years.
* Glaucomtous and nonglaucomatous participants with visually significant cataracts.
* Best-corrected visual acuity (BCVA) equal to or worse than 6/12.
* patients candidates for standard cataract surgeries without adjunctive procedure (e.g., pupil stretching or iris hooks).

Exclusion Criteria:

* Major intraoperative or postoperative complications from cataract surgery
* Peripheral anterior synechiae (PAS) detected by indentation gonioscopy.
* Uveitis, severe retinal diseases, or congenital Anomalies.
* History of ocular trauma or any intraocular Surgery. ocular trauma or any intraocular Surgery

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2019-09-20 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure change | 4 weeks
  intraocular pressure measurement by Goldman's applanation tonometr
ocular bio-metrics change | 4 weeks
  anterior chamber angle angle opening distance and anterior chamber depth change

SECONDARY OUTCOMES:
Phacoemulsification as treatment to glaucoma | 4 weeks
  intraocular pressure decrease after surgery in glaucoma patients

CONTACTS AND LOCATIONS:
Overall Officials: Karim A Raafat, MD, Study Director — Cairo University
Locations (1):
- Faculty of medicine, Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elgin U, Sen E, Simsek T, Tekin K, Yilmazbas P. Early Postoperative Effects of Cataract Surgery on Anterior Segment Parameters in Primary Open-Angle Glaucoma and Pseudoexfoliation Glaucoma. Turk J Ophthalmol. 2016 Jun;46(3):95-98. doi: 10.4274/tjo.92604. Epub 2016 Jun 6. PMID 27800269
- [Result] Melancia D, Abegao Pinto L, Marques-Neves C. Cataract surgery and intraocular pressure. Ophthalmic Res. 2015;53(3):141-8. doi: 10.1159/000377635. Epub 2015 Mar 7. PMID 25765255
- [Result] Hsu CH, Kakigi CL, Lin SC, Wang YH, Porco T, Lin SC. Lens Position Parameters as Predictors of Intraocular Pressure Reduction After Cataract Surgery in Nonglaucomatous Patients With Open Angles. Invest Ophthalmol Vis Sci. 2015 Dec 1;56(13):7807-7813. doi: 10.1167/iovs.15-17926. PMID 26650901
- [Result] Man X, Chan NC, Baig N, Kwong YY, Leung DY, Li FC, Tham CC. Anatomical effects of clear lens extraction by phacoemulsification versus trabeculectomy on anterior chamber drainage angle in primary angle-closure glaucoma (PACG) patients. Graefes Arch Clin Exp Ophthalmol. 2015 May;253(5):773-8. doi: 10.1007/s00417-015-2936-z. Epub 2015 Feb 3. PMID 25644619

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-09-14): https://cdn.clinicaltrials.gov/large-docs/73/NCT04334473/Prot_SAP_000.pdf
  • Informed Consent Form (2019-09-14): https://cdn.clinicaltrials.gov/large-docs/73/NCT04334473/ICF_001.pdf